CLINICAL TRIAL: NCT05196282
Title: An Open-label, 6-arm Parallel Group, Single-center Preference Clinical Study on the Effects of Smoking Cessation or Switching From Cigarette Smoking to the Tobacco Heating System (THS) in Adult Smokers Who Have Been Diagnosed With Inflammatory Bowel Disease (IBD) and Are Under Treatment.
Brief Title: Influence of Smoking Cessation or Switching to THS on Disease Activity in IBD Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaFCED e.K. (Other)
Responsible Party: Sponsor
Other Study IDs: HW-001-DE
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Smoking in IBD Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- UC, Smoker
  Interventions: Other: Smoking cessation
- UC, Smoking cessation
  Interventions: Other: Smoking cessation
- UC, THS user
  Interventions: Other: Smoking cessation
- CD, Smoker
  Interventions: Other: Smoking cessation
- CD, Smoking cessation
  Interventions: Other: Smoking cessation
- CD, THS user
  Interventions: Other: Smoking cessation

INTERVENTIONS:
Other: Smoking cessation — Patients are forced to stop smoking

SUMMARY:
The main goal of this study is to evaluate the effects of smoking cessation or switching from cigarette smoking to THS (tobacco heat system) on the clinical course of UC (ulcerative colitis) and CD (Crohn´s disease) in adult smokers who were diagnosed with IBD and are under treatment.

Measures using validated/standardized assessment methods and self-reported outcomes will be assessed in patients who stop smoking or switch from smoking to using THS over the investigational period of 6 months, relative to smokers who continue smoking cigarettes.

ELIGIBILITY:
Inclusion criteria:

For all patients:

1. Patient has signed the ICF (Informed Consent Form) and is able to understand the information provided in the ICF. Patient can sign or not the optional ICF on long-term biobanking of samples.
2. 19 years ≤ patient's age ≤ 75 years old
3. Patients who were diagnosed with UC or CD.
4. Patient's disease activity is mild to moderate (PMS ≤ 6; CDAI: ≤ 300) and has not changed for at least the last 3 months, as judged by the Investigator. a
5. Patient is ready to comply with the study procedures (including readiness to accept smoking abstinence and/or use of THS).
6. Patient has smoked at least 5 commercially available and/or "roll your own cigarette" every day (no cigarette brand restriction) for at least the last 1 year, based on self-reporting. Smoking status will be verified based on a urinary cotinine test (i.e., cotinine ≥ 200 ng/mL). Specific to patients who prefer to continue using nicotine-containing and tobacco product after having been advised to quit smoking:
7. Not intending to quit using THS or smoking cigarettes within the next 6 months (to be checked at V2). Specific to patients who prefer to stop smoking cigarettes:
8. Any patient who is willing to attempt quitting cigarette smoking

   Exclusion criteria:

   For all patients:
9. Patients with severe disease activity (PMS > 5; CDAI > 300), as judged by the Investigator.
10. Female patients who are pregnant or breast-feeding
11. Female patients who are planning to become pregnant during the next 8 months
12. Patients with a history of recent and current alcohol and substance abuse
13. Patient is ineligible as judged by the Investigator to participate in the study for any reason (e.g., medical, psychiatric and/or social reason), including any abnormal safety laboratory values obtained at screening that are judged as clinically significant by the investigator.
14. Patient is legally incompetent, or physically or mentally incapable of giving consent (e.g., emergency situation, under guardianship, prisoners, or patients who are involuntarily incarcerated).
15. Patient with any major illness/condition or evidence of an unstable clinical condition (e. g. renal, hepatic, hematologic, gastrointestinal [except the disease under study], endocrine, cardiovascular, pulmonary, immunologic, or local active infection/infectious illness) that, in the investigator's judgment, could impact study results.
16. The patient has colorectal carcinoma or high-grade dysplasia adenoma.
17. As per the investigator's judgment, the patient has medical conditions which require or will require in the course of the study, a medical intervention (e. g. start of treatment, surgery, hospitalization), which may interfere with the study participation and/or study results.
18. Any other clinically significant medical condition, which as per the judgment of the PI would jeopardize the safety of the patient.
19. Clinically significant ECG alterations that will not allow patient to participate in the study, per Investigator's discretion

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smoking IBD patients under treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Activity Scores | 6.5 months
  partial Mayo Score, Range from 0-9. The higher the more active
Activity Scores | 6.5 months
  CDAI, Crohn's disease activity index - Range from 0-600. The higher the more active